CLINICAL TRIAL: NCT04062812
Title: Comparison of Diluted vs Concentrated Regional Citrate Anticoagulation in Continuous Renal Replacement Therapy: A Quasi-experimental Study
Brief Title: New Protocol With Diluted Citrate in Continuous Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-CIT-2019-34
Record Dates: First submitted 2019-08-06; First posted 2019-08-20 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-02

CONDITIONS: Acute Renal Failure; Dialysis; Complications; Citrate Poisoning
Keywords: sodium citrate; calcaemia; magnesium; phosphorus; ionic calcium
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Quasi-experimental design
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diluted citrate (Experimental): Initial citrate dose 3.5 mmol/L Initial calcium programmed 100% ("compensation dose") only dialysis and ratio 1:10 (blood/dialysis) No fluids in the repositioning scale
  Interventions: Other: the same citrate dosification in both types
- Concentrated citrate (Active Comparator): Initial citrate dose: 3.5 mmol/L Initial calcium dose: 1.9 mmol/L and 1:20 ratio (blood/dialysis) No convection programmed
  Interventions: Other: the same citrate dosification in both types

INTERVENTIONS:
Other: the same citrate dosification in both types — match concentrated and dilute citrate protocol

SUMMARY:
The investigators designed a monitoring and control table of a citrate treatment on a specific monitor. This is the Baxter "Prismaflex" monitor, with 8.2 software version. Dialysis bath liquids marketed by Baxter: Biphozyl are used. Citrate liquid (1:18) Regiocit is used.

The dialysis treatment monitor (CVVHD) is programmed, with a blood / citrate pumps at a rate of 1:10 (1 ml / min of blood: 10 ml / h of dialysis fluid) The starting dose of citrate will be 3.5 mmol / l and the calcium compensation will be 100% Working hypothesis: The patient undergoing citrate anticoagulation according to the designed algorithm will respond with ion stability and pH during the treatment, in addition to achieving an effective cleaning process.

DETAILED DESCRIPTION:
Study design: quasi-experimental design. two groups:

1. Usual protocol with Multifiltrate monitor and citrate (136 mmol/l)
2. Intervention group. New protocol with Prismaflex monitor and citrate (18 mmol/l)

Study population Inclusión/exclusion criteria:

Adult patients (regardless of their underlying pathology), who develop acute renal failure, admitted to the ICU of St Pau Hospital with the Intensive Medicine medical team, who require citrate anticoagulation in continuous dialysis therapy and are treated with Baxter "Prismaflex" monitor.

Patients who meet the criteria described above will be followed up in this study.

Expected sample size:

It is estimated that with 24/12 (group1/2) patients will be enough to achieve our goal

Methodology. Information sources:

The start of the treatment with Baxter citrate will be given according to the patient's need and subject to a basic medical decision. From here the research team will enter. The investigation team will never influence the medical decision.

Since such a treatment is started, the main investigator will assign a number to the dialysis circuit and will be followed, every six hours, for the most important variables. The rest of the variables will be collected at least once a day and according to the patient's situation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (regardless of their underlying pathology), who develop acute renal failure, admitted to the ICU of St Pau with the medical team of Intensive Medicine, who require anticoagulation with citrate in continuous dialysis therapy and are treated with the Baxter monitor.

Exclusion Criteria:

* parenteral nutrition
* pregnancy
* cardiac surgery
* coronary patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Dialysis flow | 6 hours
  Speed at which the dialysis fluid pump is programmed in the circuit and measured in milliliters / hour
Blood flow | 6 hours
  Speed at which the blood pump is programmed in the dialysis circuit and measured in milliliters / min
Citrate dose | 6 hours
  Relationship that exists between the liquid we infuse (which contains 18mmol / L citrate) and the blood pump. It is measured in mmol citrate / liter of blood
Calcium dose | 6 hours
  Amount of calcium that is replenished to the patient when the dialyzed blood is returned. It is measured in%.

SECONDARY OUTCOMES:
Filter operating hours | number of hours
  They correspond to the hours that go from the beginning of the circuit until the end of the circuit in which the fungible is discarded. It can be several days
Arterial pH | 6 hours
  Corresponds to the patient's arterial blood pH figure at the time of observation
Arterial bicarbonate | 6 hours
  It is the bicarbonate figure found in arterial blood. It is measured in mmol / l.
Post-filter ionic calcium | 6 hours
  Corresponds to the value of ionic calcium by taking the sample at the blood outlet of the dialysis filter. It is measured in mmol / l.
Ionic Calcium Patien | 6 hours
  It is the ionic calcium value of the patient in a systemic way, preferably arterial. It is measured in mmol / l
Total calcium | 6 hours
  Total calcium value. It is measured in mmol / l
Total Ca / Ionic Ca Ratio | 24 hours
  Relationship between the total calcium and the ionic one of the patient
Match | 24 hours
  Value of this ion in the patient. It is measured in mmol / l.
Magnesium | 24 hours
  Value of this ion in the patient. It is measured in mmol / l.
Sodium | 24 hours
  Value of this ion in the patient. It is measured in mmol / l.
Potassium | 24 hours
  Value of this ion in the patient. It is measured in mmol / l.
Urea | 24 hours
  Urea level of the patient at the time of observation
Creatinine | 24 hours
  Creatinine level of the patient at the time of observation
INR | 24 hours
  INR level of the patient at the time of observation
Lactate | 24 hours
  Lactate level of the patient at the time of observation

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació de Gestió Sanitària de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Spain